CLINICAL TRIAL: NCT03508388
Title: Prognostic Value of Liver Volume on Acute Decompensation of Alcoholic Cirrhosis, a Prospective Multicenter Observational Study
Brief Title: Value on Survival of Liver Volume After an Acute Decompensation of an Alcoholic Cirrhosis
Acronym: PROLIV
Status: Terminated | Type: Observational
Why Stopped: inclusion number not sufficient
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Nīmes (Unknown); Narbonne Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0022
Record Dates: First submitted 2018-04-23; First posted 2018-04-25 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2020-01

CONDITIONS: Alcoholic Cirrhosis; Alcoholic Liver Disease
Keywords: Liver volume; Alcoholic cirrhosis; Liver transplantation
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Liver Diseases, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigator seek to determine whether the volume of the liver can predict the survival after a decompensation of a patient suffering from chronic liver disease caused by excessive alcohol consumption (or alcoholic cirrhosis). Our hypothesis is that patients with a "small" liver have a lower survival compared to patients having a "normal" sized liver.

DETAILED DESCRIPTION:
In this observational, prospective and multicentre clinical trial, investigator seek to determine the prognostic value of liver volume during an acute decompensation. Investigator plan to enroll admitted adult patients with acute decompensation of an alcoholic cirrhosis (abstinent or not), followed for one year or until death or liver transplantation. Liver volume will be evaluated using CT-scan or MRI reconstructions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patient suffering from alcoholic cirrhosis (withdrawn or not)
* Patient admitted in emergency for an alcoholic cirrhosis decompensation only
* Prescription for a cutting imaging (CT scan or MRI) during hospitalisation
* Alcohol consumption of more than 3 units per day for men and 2 units for women in average, over at least the last 5 years before the cirrhosis diagnosis
* Patient suffering from decompensated cirrhosis defined by at least one of the following criteria : Model For End-Stage Liver Disease (MELD) score above or equal to 15, ascites needing iterative punctures, symptomatic bacterial ou fungal infections, acute digestive bleeding due to portal hypertension, hepatic encephalopathy defined by a West Haven score above or equal to 2

Exclusion Criteria:

* Nodule with typical criteria of hepatocellular carcinoma
* B or C viral infections actives
* Presence of transjugular intrahepatic portosystemic shunt (TIPS)
* Presence of an occlusive thrombosis of the porta or one of the principal branches
* Presence of a thrombosis of the sus-hepatic vein
* Active extra-hepatic malignant tumor
* Decompensated cardio-vascular disease
* Patient unwilling to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from alcoholic cirrhosis, withdrawn or not, hospitalised for an acute decompensation
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
All cause mortality or liver transplantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jose URSIC BEDOYA, MD, Principal Investigator — UH Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No